CLINICAL TRIAL: NCT02040285
Title: Low-dose Laxative Improves Performance and Feasibility of Computed Tomography Colonography (CTC). Comparison vs Laxative Free CTC.
Brief Title: Low-dose Laxative Improves Performance and Feasibility of Computed Tomography Colonography (CTC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Andrea Laghi, Prof., MD, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTC-Prep 1
Record Dates: First submitted 2014-01-13; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Gastrointestinal Complication
Keywords: CT colonography
MeSH Terms: interventions — Bisacodyl; Iopamidol

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Free laxative CTC (Active Comparator)
  Interventions: Drug: Iopamidol
- Low-dose laxative bowel preparation for CTC (Experimental)
  Interventions: Drug: Bisacodyl & PEG-CS

INTERVENTIONS:
Drug: Bisacodyl & PEG-CS — the day before the CTC:
  * low fiber diet
  * at 15.00: 2 tablets of bisacodyl (5 mg)
  * at 17.00: 1 litre of PEG-CS
  * liquid diet
  the day of the exam:
  * at home: 2 tablets of bisacodyl (5 mg)
  * at the Hospital (3 hours after tablets intake): 90 ml of Iopamidol in 500 ml of water
  * at the Hospital (5 minutes after Iopamidol intake): 10 mg of Metoclopramide mono chlorohydrate monohydrate im
  Other Names: Lovoldyl (Bisacodyl); Lovolesse (PEG-CS); Gastromiro (Iopamidol); Plasil (Metoclopramide mono chlorohydrate monohydrate)
  Arms: Low-dose laxative bowel preparation for CTC
Drug: Iopamidol — the day before CTC:
  * low fiber diet
  * at 15.00: 90 ml of Iopamidol in 250 ml of water
  * at 17.00: 90 ml of Iopamidol in 250 ml of water
  * at 20.00: start liquid diet
  Other Names: Gastromiro (Iopamidol)
  Arms: Free laxative CTC

SUMMARY:
The aim of this study is to evaluate a low-dose of bowel preparation for Computed Tomography Colonography (CTC) versus free laxative CTC with regard to performance, feasibility, patient tolerability and acceptance.

DETAILED DESCRIPTION:
Computed Tomography Colonography (CTC) is a valid alternative to colonoscopy in the detection of cancer, polyps and other colon lesions.

High volume cathartic preparations, low volume cathartic solutions with oral tagging agent and tagging agent only are the procedures available for CTC.

High volume preparations are a considerable burden for patients. Low volume cathartic solutions are more accepted by the patients, reduce the amount of tagging agent and the waiting time to the exam. Tagging agent only preparations represent a risk if they are taken without medical supervision.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients undergoing a CTC
* Patient written informed consent

Exclusion Criteria:

* Pregnant or lactating women or at a risk of becoming pregnant
* Known or suspected gastrointestinal obstruction or perforation, toxic megacolon, ileo, major colonic surgery
* History of anaphylaxis to Iopamidol or allergic reactions to drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Efficacy | 20 min
  Tagging. In prone and supine position, each colon segment (caecum, ascending, transverse, descending, sigma and rectum) will be graded by using a 4 point scale (from 0= greater than 75% of residuals to 3= minor than 25% of residuals).

SECONDARY OUTCOMES:
Efficacy | 20 minutes
  Residual fluid evaluation. In prone and supine position, each colon segment (caecum, ascending, transverse, descending, sigma and rectum) will be graded by using a 4 point scale (from 1= minor than 25% of the ap axis to 4= greater than 75% of the ap axis).
Efficacy | 20 min
  Bowel distension. In prone and supine position, each colon segment (caecum, ascending, transverse, descending, sigma and rectum) will be graded by using a 4 point scale (from 0= greater than 75% of the maximal distension to 3= minor than 25% of the maximal distension)
Safety | 2 days (the day before and the day of CTC)
  Recording of all Adverse Events (AEs) occurring during the 2 days of treatment
Safety | 2 days (the day before and the day of the exam)
  Tolerability. Recording of gastrointestinal (GI) symptoms occurring during the 2 days of treatment. Intensity of GI symptoms will be evaluated by a Visual Analgic Scale (VAS) ranging from 0=no symptoms to 10=severe, as much as possible.
Acceptability | 2 days (the day before and the day of the exam)
  Evaluation of the patient discomfort related to bowel preparation. A 4 point scale is used: 1=none; 2=mild distress; 3=moderate distress; 4=severe distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Umberto I, Roma, Italy